CLINICAL TRIAL: NCT00843297
Title: Clinical and Neurological Outcome With Two Different Cooling Methods (Invasive and Non-invasive) After Sudden Cardiac Arrest
Brief Title: COOL-Trial: Outcome With Invasive and Non-invasive Cooling After Cardiac Arrest
Acronym: COOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Holger Thiele, Assistant Professor, University of Leipzig, Heart Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: COOL-Trial
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Cardiac Arrest; Hypothermia
Keywords: Sudden Cardiac Arrest; Hypothermia; Outcome, neurological; Coolgard; ArcticSun
MeSH Terms: conditions — Heart Arrest; Hypothermia; Death, Sudden, Cardiac; Neurologic Manifestations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- CG (Active Comparator): Coolgard: invasive Cooling
  Interventions: Device: Coolgard
- AS (Active Comparator): ArcticSun: Surface-Cooling
  Interventions: Device: ArcticSun
- UnCOOL (Sham Comparator): No Cooling-Therapy due to non-operational cooling-devices
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Device: Coolgard — invasive Cooling via femoral ICY-catheter
  Arms: CG
Device: ArcticSun — Noninvasive surface-cooling by saline-cooled thermo-vest
  Arms: AS
Other: Conventional treatment — Intensive care-treatment without cooling
  Arms: UnCOOL

SUMMARY:
Sudden cardiac arrest (SCA) remains one of the major leading causes of death. Cognitive deficits are common in survivors of SCA. Postresuscitative mild induced hypothermia (MIH) lowers mortality and reduces neurologic damage after cardiac arrest. The investigators evaluated the efficacy and side effects of therapeutic hypothermia in an unselected group of patients after SCA.

DETAILED DESCRIPTION:
Consecutive patients with restoration of spontaneous circulation (ROSC) after resuscitation due to out-of-hospital SCA, admitted to our intensive care unit, underwent MIH. Hypothermia was induced by infusion of cold saline and whole-body-cooling methods (electronic randomization: invasive Coolgard or non-invasive ArcticSun). The core body temperature was operated at 32 to 34 °C over a period of 24 hours followed by active rewarming. Neurological status was evaluated at hospital discharge and 6 months after discharge using the Pittsburgh Cerebral Performance Category (CPC). Blood samples of neuron-specific enolase (NSE) were collected during 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* ROSC after SCA due to VF/VT or PEA/Asystolia
* GCS 3

Exclusion Criteria:

* Non-cardiac SCA
* Pregnancy
* Unstable Circulation instead of High-dose Inotropics
* Life-expectancy reducing concomitant illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Time to reach the target temperature | Twenty-four hours
NSE as a parameter for cerebral damage | Seventy-two hours

SECONDARY OUTCOMES:
Neurologic outcome | Six months
Survival | Six months
Periprocedural complications | Seventy-two hours

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, Associate Professor, Principal Investigator — Study Chair; Undine Pittl, MD, Study Director — Study Sub-Investigator
Locations (1):
- University of Leipzig, Heart Center, Cardiology, Leipzig, Germany

REFERENCES:
- [Background] Zeiner A, Holzer M, Sterz F, Behringer W, Schorkhuber W, Mullner M, Frass M, Siostrzonek P, Ratheiser K, Kaff A, Laggner AN. Mild resuscitative hypothermia to improve neurological outcome after cardiac arrest. A clinical feasibility trial. Hypothermia After Cardiac Arrest (HACA) Study Group. Stroke. 2000 Jan;31(1):86-94. doi: 10.1161/01.str.31.1.86. PMID 10625721
- [Background] Bernard SA, Gray TW, Buist MD, Jones BM, Silvester W, Gutteridge G, Smith K. Treatment of comatose survivors of out-of-hospital cardiac arrest with induced hypothermia. N Engl J Med. 2002 Feb 21;346(8):557-63. doi: 10.1056/NEJMoa003289. PMID 11856794